CLINICAL TRIAL: NCT02325726
Title: Renal Resistive Index Compared With NephroCheckTM to Predict Postoperative Acute Renal Failure in Patients Undergoing Cardiac Surgery.
Brief Title: RRI Compared With NephroCheckTM to Predict Acute Renal Failure After Cardiac Surgery.
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX RNI 02/2014
Record Dates: First submitted 2014-12-21; First posted 2014-12-25 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Cardiac Surgery; Extracorporeal Circulation; Nephrocheck; Renal Failure
Keywords: Cardiac surgery; Extracorporeal circulation; Renal failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal Resistive Index/Nephrocheck test: Patients undergoing elective cardiac surgery with extracorporeal circulation and who are at risk to develop postoperative Acute Kidney Injury.
  Interventions: Procedure: Renal Resistive Index compared with NephroCheckTM

INTERVENTIONS:
Procedure: Renal Resistive Index compared with NephroCheckTM

SUMMARY:
Postoperative acute renal failure is a frequent complication after cardiac surgery. The current practice cannot predict Acute Kidney Injuries (AKI) early enough to reduce a significant kidney assault and prevent an organic dysfunction leading to cortical tubular necrosis.

Several recent studies in cardiac surgery have shown that, both sonographic criteria, such as the Renal Resistive Index (IRR) and urinary biomarkers can predict AKI promptly. These urinary biomarkers are the 'tissue inhibitor of metalloproteinases' (TIMP-2) and the 'insulin-like growth factor binding protein' (IGFBP7). These two proteins are sought noninvasively, directly in the urine, within the same test called 'NephroCheckTM'. These markers, ultrasonographic and biologic, have the advantage of being easy to perform, accessible and seem to have both high sensitivity and specificity to predict AKI promptly after cardiac surgery. Thus, the IRR and the NephroCheckTM test could become essential tests to guide clinicians in determining rapidly whether a patient will develop AKI. However, so far, no study has compared these markers yet.

Therefore, the aim of this prospective observational study will be to compare the effectiveness of the IRR with the NephroCheckTM to predict AKI promptly after cardiac surgery. The secondary outcome will be to determine the threshold of these markers from which patients will be likely to develop AKI

ELIGIBILITY:
Inclusion Criteria:

* Elective patients
* Patients scheduled to receive an extracorporeal circulation
* Patients aged 60 and older
* Patients at risk of postoperative acute kidney injury presenting at least two of the following risk factors:

  * Age > 60 years.
  * Arteritis defined as severe lower limb arteriopathy or carotid stenosis > 50%
  * Diabetes
  * Valvular or combined surgery
  * Preoperative intra-aortic balloon pump.

Exclusion Criteria:

* Unable to provide informed consent
* Comatose patients
* Patients with dementia
* Patient who underwent a previous sternotomy
* Chronic renal failure (sCr clearance < 30 ml.min-1)
* Renal artery stenosis
* Endocarditis
* Emergent surgery
* Nephrotoxic treatment
* Non-sinus cardiac rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery with extracorporeal circulation and who are at risk to develop postoperative Acute Kidney Injury.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Renal Resistive Index compared with NephroCheckTM | Day 0 (inclusion) / after cardiac surgery
  Compare the effectiveness of the IRR with the NephroCheckTM to predict AKI after cardiac surgery. AKI will be defined according to the RIFLE criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Cédrick ZAOUTER, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Pessac, Bordeaux, France